CLINICAL TRIAL: NCT03757533
Title: Health Coaching as a Tool for Improving Medication Adherence in Adult Patients With Inflammatory Bowel Disease: A Prospective Randomized Study
Brief Title: Health Coaching as a Tool for Improving Medication Adherence in Adult Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Sara Horst, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 182030
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Coaching (Experimental): Participants in the Health Coaching (HC) arm will be assigned to a health coach for a period of 5 months along with receiving usual care (UC). An initial telephone call with the coach will include a discussion about the participant's self-assessment of health perceptions and goals. This self-assessment creates the foundation for the personalization of the behavioral intervention. From this point, the participant schedules the remaining 9 biweekly sessions (30-45 minute in length), for a total of 10 coaching calls over 5 months. Sociodemographic, behavioral, and psychosocial data will be collected over a period of 24 months by surveys and from the medical record.
  Interventions: Behavioral: Health Coaching; Other: Surveys
- Control (Other): Participants in the control arm will receive usual care (UC). Sociodemographic, behavioral, and psychosocial data will be collected over a period of 24 months by surveys and from the medical record. To enhance recruitment, those subjects randomized to the usual care control group will be offered to participate in the health coaching arm of the study as well after a period of 6 months. If they refuse, they will continue in the usual care control group.
  Interventions: Other: Surveys

INTERVENTIONS:
Behavioral: Health Coaching — 10 phone calls with a trained health coach
  Arms: Health Coaching
Other: Surveys — Surveys to assess Behavioural and Psychosocial measures

SUMMARY:
Inflammatory bowel disease (IBD) including Crohn's disease (CD) and Ulcerative colitis (UC) is a chronic idiopathic intestinal disorder involving the interplay of environmental, immunomodulatory and genetic causative factors. Treatment for IBD is multimodal and includes lifestyle modification, chronic pharmacotherapy and surgery. Given the need for chronic pharmacotherapy, medication adherence is a crucial therapeutic goal in the management of IBD. In fact, medication non-adherence has been associated with greater risk of relapse and increased healthcare costs.

In a previous study, the investigators found clinically identifiable risk factors for non-adherence for self-injectable biologic medications in a population with moderate to severe CD. These risk factors included smoking, prior biologic use, psychiatric history, and current narcotic use. The primary objective of this study is to use a multidisciplinary team approach that implements a targeted coaching intervention to promote behavioral change and improve medication adherence in adult patients with IBD who are at high risk of non-adherence.

ELIGIBILITY:
Inclusion Criteria:

* adult patients treated at the Inflammatory Bowel Disease (IBD) clinic at Vanderbilt with Crohn's disease or Ulcerative colitis confirmed by endoscopy or radiology assessment
* currently prescribed a biologic agent (self-injectable or infusion) for management of IBD
* medication dispensing is documented in patient medical record

Exclusion Criteria:

* patients less than 18 years of age
* unstable clinical condition (bleeding, infection, intestinal obstruction, etc.)
* patients who are required to get biologic medication at a specialty pharmacy outside of Vanderbilt University that is not documented in medical record(exclusion due to inability to accurately track prescription refills)
* patients with short bowel syndrome, an ostomy, obstructive disease with strictures, history of tuberculosis, hypersensitivity reaction to anti-TNF agent, cancer, renal failure requiring specific treatment such as dialysis
* patients with severe psychological comorbidity, defined as reported intent to self-harm or harm others or psychiatric hospitalization in the past year
* patients with current alcohol abuse or illegal drug use ascertained by medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Medication Adherence MPR | 24 months
  Medication adherence will be measured using the medication possession ratio (MPR). MPR is calculated as the sum of days' supply for all prescription claims divided by the total number of days elapsed during that period.
Medication Adherence PDC | 24 months
  Medication adherence will be measured using the proportion of days covered (PDC). PDC is calculated as the number of days the patient has medication divided by the total number of days elapsed during that period.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Horst, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center Inflammatory Bowel Disease Clinic, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391